CLINICAL TRIAL: NCT07396402
Title: Study of Scube-1 and Scube-3 in Polycystic Ovary Syndrome (PCOS) and Their Possible Use as Inflammatory Markers and as a Link Between PCOS and Cardiovascular Events.
Brief Title: SCUBE Proteins in Polycystic Ovary Syndrome (IPSOS)
Acronym: IPSOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7725
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Insulin Resistance
Keywords: SCUBE-1; SCUBE-3; Polycystic Ovary Syndrome; PCOS; Insulin Resistance; Inflammation; Cardiovascular Risk
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: PCOS - Normoinsulinemic (Experimental): Description: Women with PCOS and normal insulin sensitivity Intervention: Blood sample collection for SCUBE-1 and SCUBE-3 measurement by ELISA
  Interventions: Diagnostic Test: Blood Sample Collection for SCUBE-1 and SCUBE-3 Measurement
- Arm 2: PCOS - Hyperinsulinemic (Experimental): Description: Women with PCOS and insulin resistance Intervention: Blood sample collection for SCUBE-1 and SCUBE-3 measurement by ELISA
  Interventions: Diagnostic Test: Blood Sample Collection for SCUBE-1 and SCUBE-3 Measurement
- Arm 3: Healthy Controls (Experimental): Description: Healthy women of reproductive age without PCOS Intervention: Blood sample collection for SCUBE-1 and SCUBE-3 measurement by ELISA
  Interventions: Diagnostic Test: Blood Sample Collection for SCUBE-1 and SCUBE-3 Measurement

INTERVENTIONS:
Diagnostic Test: Blood Sample Collection for SCUBE-1 and SCUBE-3 Measurement — Blood sample collection performed specifically for research purposes to measure circulating SCUBE-1 and SCUBE-3 levels using enzyme-linked immunosorbent assay (ELISA).

SUMMARY:
This study investigates circulating levels of SCUBE-1 and SCUBE-3 proteins in women with polycystic ovary syndrome (PCOS) compared with healthy controls. Differences between normoinsulinemic and hyperinsulinemic PCOS subgroups will be evaluated, as well as correlations with clinical and metabolic parameters related to inflammation and cardiovascular risk.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age and is frequently associated with insulin resistance, chronic low-grade inflammation, and increased cardiovascular risk.

SCUBE proteins (Signal peptide-CUB-EGF domain-containing proteins) are recently identified molecules involved in inflammation, angiogenesis, and platelet activation. Their role in PCOS has not been fully elucidated.

This interventional, non-randomized study will measure circulating SCUBE-1 and SCUBE-3 levels in women with PCOS and healthy controls. PCOS patients will be stratified into normoinsulinemic and hyperinsulinemic subgroups based on previously performed metabolic assessments. Blood samples will be collected during routine clinical practice and analyzed using ELISA assays. The study aims to assess SCUBE proteins as potential biomarkers of inflammation and cardiovascular risk in PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18-35 years
* Diagnosis of polycystic ovary syndrome (normoinsulinemic or hyperinsulinemic)
* Availability of basal hormonal evaluation and oral glucose tolerance test
* Healthy women for control group
* Written informed consent

Exclusion Criteria:

* Pregnancy
* History of cardiovascular disease
* Diabetes mellitus or impaired glucose tolerance
* Hypertension
* Significant hepatic or renal disease
* Other endocrine disorders
* Neoplastic diseases
* Psychiatric disorders
* Autoimmune diseases
* Shift work
* Obesity
* Refusal to sign informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Circulating SCUBE-1 levels | At enrollment
  Comparison of SCUBE-1 plasma concentrations among normoinsulinemic PCOS, hyperinsulinemic PCOS, and healthy controls

SECONDARY OUTCOMES:
Circulating SCUBE-3 levels | At enrollment
  Comparison of SCUBE-3 plasma concentrations among study groups
Correlation with clinical and laboratory parameters | At enrollment
  Association between SCUBE-1 and SCUBE-3 levels and clinical (age, BMI, hirsutism, acne, menstrual irregularities) and laboratory variables (lipid profile, androgen levels)

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Apa, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No